CLINICAL TRIAL: NCT00746603
Title: A Feasibility Study to Evaluate the Safety of Simvastatin in Young Adults Treated for Hodgkin's Disease
Brief Title: Feasibility Study of Simvastatin in Hodgkin's Lymphoma Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAB4447
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A Intervention Arm (Experimental): Escalating dose of simvastatin in subjects who are survivors of Hodgkin Lymphoma
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — All patients will start at 10mg of simvastatin, and then, based on results of interim evaluation escalated to 20mg and then 40. Patients will stay on maximally tolerated dose of drug until the end of the study at 26 weeks.
  Other Names: Zocor

SUMMARY:
Lay abstract: Study Purpose With contemporary combined modality therapy the expected longterm survival of children and adolescents with Hodgkin's disease (HD) is exceedingly high. Thus, the emphasis for future therapeutic interventions must include attention to the late effects of therapy. The development of cardiovascular disease as a late effect of radiation therapy has been well described and documented. Our recent pilot study of child and young adult HD survivors revealed significant subclinical atherosclerosis as evidenced by increased Carotid Artery Intima Media Thickness (CIMT) compared to controls. The higher CIMT values were positively associated with increasing age, total cholesterol, LDLcholesterol and diastolic BP. This finding was present in children and young adults who had received no or low dose radiation suggesting that chemotherapy or the disease process itself contributes to the development of atherosclerosis and risk for cardiovascular disease. Numerous studies have shown HMG CoA reductase inhibitors ("statins") to be effective in reducing the progression of atherosclerosis in adults. These agents have been studied in children and young adults for over a decade.

The primary aim of this study is:

To obtain pilot safety data on the use of simvastatin in young adults treated for HD.

The secondary aims of this study are:

To obtain pilot data on the effect of simvastatin on subclinical carotid artery atherosclerosis as measured by Carotid Artery IMT in young adults treated for HD.

To obtain pilot data on the effect of simvastatin on markers of inflammation measured in the serum of young adults treated for HD.

To obtain pilot data to serve as the basis for the development of a multicenter randomized study for the use of simvastatin in survivors of HD.

DETAILED DESCRIPTION:
With contemporary combined modality therapy the expected longterm survival of children and adolescents with Hodgkin's disease (HD) is exceedingly high. Thus, the emphasis for future therapeutic interventions must include attention to the late effects of therapy. The development of cardiovascular disease as a late effect of radiation therapy has been well described and documented. Our recent pilot study of child and young adult HD survivors revealed significant subclinical atherosclerosis as evidenced by increased Carotid Artery Intima Media Thickness (CIMT) compared to controls. The higher CIMT values were positively associated with increasing age, total cholesterol, LDLcholesterol and diastolic BP. This finding was present in children and young adults who had received no or low dose radiation suggesting that chemotherapy or the disease process itself contributes to the development of atherosclerosis and risk for cardiovascular disease. Numerous studies have shown HMG CoA reductase inhibitors ("statins") to be effective in reducing the progression of atherosclerosis in adults. These agents have been studied in children and young adults for over a decade.

The primary aim of this study is:

To obtain pilot safety data on the use of simvastatin in young adults treated for HD.

The secondary aims of this study are:

To obtain pilot data on the effect of simvastatin on subclinical carotid artery atherosclerosis as measured by Carotid Artery IMT in young adults treated for HD.

To obtain pilot data on the effect of simvastatin on markers of inflammation measured in the serum of young adults treated for HD.

To obtain pilot data to serve as the basis for the development of a multicenter randomized study for the use of simvastatin in survivors of HD.

We will do this by enrolling patients diagnosed with HD and evaluating the safety of simvastatin as evidenced by laboratory measures

ELIGIBILITY:
Inclusion Criteria:

* At least three years from completion of treatment for Hodgkin's Disease
* Age 18- 35
* Ability to complete self report questionnaires in either English or Spanish
* Willingness of patient, or parent/guardian if patient less than 18 years of age to sign consent to participate in study
* Willingness of patient to sign assent if greater than 7 years of age and less than 18 years

Exclusion Criteria:

* Pregnant or breast feeding
* Tanner Stage 1
* Currently taking cyclosporine, niacin, antiretrovirals, macrolide antibiotic, azole antifungal
* Liver enzymes greater than 1.5 times the upper level of normal
* Creatine Kinase greater than 2 times the upper level of normal
* Use of estrogen containing contraceptive

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Levine, MD, Principal Investigator — Columbia Univeristy Medical Center
Locations (1):
- Columbia Univeristy Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment occurred in the late effects clinic
Groups:
- Simvastatin: Escalating dose of simvastatin
  Simvastatin: All patients will start at 10mg of simvastatin, and then, based on results of interim evaluation escalated to 20mg and then 40. Patients will stay on maximally tolerated dose of drug until the end of the study at 26 weeks.
Period: Overall Study
Arm/Group | Simvastatin
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Simvastatin
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Grade 3 or Greater Muscle Toxicity
Description: Number of participants experiencing grade 3 or greater muscle toxicity as evaluated by creatinine kinase laboratory tests.
Time Frame: Up to 26 weeks
Population: The study terminated in 2009 due to poor enrollment. The principal investigator (PI) and study team are no longer at the institution and the PI has confirmed that the data no longer exists. There are no data to report.
Arm/Group | Simvastatin
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants Experiencing Grade 3 or Higher Liver Toxicity
Description: Number of participants experiencing grade 3 or higher liver toxicity as determined by liver function laboratory tests.
Time Frame: Up to 26 Weeks
Population: as for outcome 1
Arm/Group | Simvastatin
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Carotid Intima-media Thickness Test (CIMT)
Description: A change in CIMT measurements ( measured in millimeters (mm)) will be performed.
Time Frame: Up to 26 Weeks
Population: as for outcome 1
Arm/Group | Simvastatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=3)
Creatine Kinase (Musculoskeletal and connective tissue disorders) | 1 (1) — S #1 at CHOP had increased CK:did not meet adverse event criteria. Later admitted to taking Androgel, not a study exclusion criteria but similar to a drug that was. PI at CHOP made decision to remove patient from study. Repeat CK wnl.
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — S#2 at CHOP developed rash, chose to stop taking medication.

LIMITATIONS AND CAVEATS:
Early termination due to poor accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes